CLINICAL TRIAL: NCT06202391
Title: Autogenic Inhibition Versus Reciprocal Inhibition Muscle Energy Techniques Effect on Swimming Performance on Swimmers With Scapular Dyskinesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/27
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Scapular Dyskinesis
Keywords: Scapular Dyskinesis, Autogenic inhibition, Reciprocal inhibition, Muscle energy Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Autogenic inhibition muscle energy technique) (Experimental): 12 sessions will be conducted over a period of 4 weeks with 3 days per week Frequency: 12 sessions, four times a week for 3 consecutive weeks Time duration: apporx. 8 to 10 minutes
  Interventions: Procedure: Autogenic Inhibition-MET
- Group B (Reciprocal inhibition muscle energy technique) (Experimental): 12 sessions will be conducted over a period of 3 weeks with 4 days per week
  Frequency: 12 sessions, four times a week for 3 consecutive weeks Time duration: apporx. 8 to 10 minutes
  Interventions: Procedure: Reciprocal Inhibition-MET protocol

INTERVENTIONS:
Procedure: Autogenic Inhibition-MET — Autogenic Inhibition-MET protocol: 3-5 repetitions of post isometric relaxation (PIR) (30- 50% isometric contraction of the muscle to be stretched for 5-10 seconds, followed by rest period of 5 seconds and then a stretch of 20-30 seconds' hold. A total of 12 sessions, four times a week, for three consecutive weeks.
  Arms: Group A (Autogenic inhibition muscle energy technique)
Procedure: Reciprocal Inhibition-MET protocol — Reciprocal Inhibition-MET protocol: 3-5 repetitions of Reciprocal Inhibition (RI) MET (30- 50% isometric contraction of the muscle opposite to the muscle to be stretched for 5-10 seconds, followed by rest period of 5 seconds and then a stretch of 20-30 seconds' hold A total of 12 sessions, four times a week, for three consecutive weeks
  Arms: Group B (Reciprocal inhibition muscle energy technique)

SUMMARY:
Swimming can cause shoulder pain due to scapular dyskinesis. Proper scapula movement is necessary for efficient swimming strokes and to avoid injury. Studying the effects of autogenic and reciprocal inhibition muscle energy techniques on swimmers with scapular dyskinesis can lead to effective interventions and reduce shoulder injuries

DETAILED DESCRIPTION:
Efficient swimming strokes require proper positioning of the scapula. Scapular dyskinesis (SD) is a condition where normal scapular kinematics are altered due to injury or changes in muscle activation. Swimmers, who are considered overhead athletes, have risk of developing SD. Even individuals who do not experience symptoms can have SD, and it may lead to future shoulder injuries. Early diagnosis and treatment of this condition can prevent it from progressing and minimize the risk of injury. Additionally, using autogenic and reciprocal inhibition muscle energy techniques can enhance the activation of the appropriate muscles responsible for scapular movement, which can lead to more effective interventions, improved swimming performance, and reduced injury risk. he intervention protocol (Muscle energy techniques to the upper fibers of the Trapezius, Levator Scapulae, Pectoralis Major, Latissimus Dorsi) will be conducted for 8-14 minutes over 3 weeks with 12 sessions/4 times a week. Outcomes measure will be assessed after the intervention period and data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Swimmers with at least four times training per week
* Does not have any shoulder pain or injury or operation to the shoulders
* Positive Scapular Dyskinesis diagnosis test
* Freestyle (also known as a front crawl) swimming stroke

Exclusion criteria:

* Shoulder pain in the last six months
* History of shoulder surgery or fracture within the last six months
* Frequent practice of physical activity in any other sport
* Negative result of the Scapular Dyskinesis test
* Other swimming strokes

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Stroke velocity | 3 weeks
  Stroke velocity will be assessed using KINOVEA
Stroke rate | 3 weeks
  Stroke rate will be assessed using KINOVEA
stroke length | 3 weeks
  Stroke length will be assessed using KINOVEA
Total strokes | 03 Week
  Total strokes will be assessed using KINOVEA
Stroke time | 03 Week
  Stroke time will be assessed using KINOVEA

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan